CLINICAL TRIAL: NCT06907173
Title: Ketamine add-on Therapy for Established Status Epilepticus Treatment Trial (KESETT)
Acronym: KESETT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: University of Michigan (Other); Medical University of South Carolina (Other); Massachusetts General Hospital (Other); Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Jaideep Kapur, MD, Eugene Meyer III Professor of Neuroscience and Professor of Neurology, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSR231657
Record Dates: First submitted 2025-03-24; First posted 2025-04-02 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Status Epilepticus
MeSH Terms: conditions — Status Epilepticus | interventions — Levetiracetam; Levamisole; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Levetiracetam (Active Comparator): Levetiracetam (LEV) (60 mg/Kg)
  Interventions: Drug: Levetiracetam (LEV) (60 mg/Kg)
- Levetiracetam + low dose Ketamine (Experimental): LEV 60 mg/mL + 1 mg/mL KET
  Interventions: Drug: Levetiracetam (LEV) (60 mg/Kg) + 1 mg/kg Ketamine (KET)
- Levetiracetam + high dose Ketamine (Experimental): LEV 60 mg/mL + 3 mg/mL KET increasing up to a weight of 75 kg
  Interventions: Drug: Levetiracetam (LEV) (60 mg/Kg) + 3 mg/kg Ketamine (KET)

INTERVENTIONS:
Drug: Levetiracetam (LEV) (60 mg/Kg) + 1 mg/kg Ketamine (KET) — The study drug will be produced at the central pharmacy, a GMP facility at the University of California, Davis. Diluted formulations are expected to remain stable for months when stored at room temperature. Expiration dates for study drugs will be determined and adjusted based on ongoing stability testing performed on study drugs prepared at the GMP facility for the study.
  All three formulations will be transparent solutions. None of the formulations are reported to consistently cause adverse effects at the infusion site. The method of drug administration, including volume and rate of infusion, is identical for all three drugs. These factors ensure that drug administration will be blinded.
  Arms: Levetiracetam + low dose Ketamine
Drug: Levetiracetam (LEV) (60 mg/Kg) + 3 mg/kg Ketamine (KET) — The study drug will be produced at the central pharmacy, a GMP facility at the University of California, Davis. Diluted formulations are expected to remain stable for months when stored at room temperature. Expiration dates for study drugs will be determined and adjusted based on ongoing stability testing performed on study drugs prepared at the GMP facility for the study.
  All three formulations will be transparent solutions. None of the formulations are reported to consistently cause adverse effects at the infusion site. The method of drug administration, including volume and rate of infusion, is identical for all three drugs. These factors ensure that drug administration will be blinded.
  Arms: Levetiracetam + high dose Ketamine
Drug: Levetiracetam (LEV) (60 mg/Kg) — The study drug will be produced at the central pharmacy, a GMP facility at the University of California, Davis. Diluted formulations are expected to remain stable for months when stored at room temperature. Expiration dates for study drugs will be determined and adjusted based on ongoing stability testing performed on study drugs prepared at the GMP facility for the study.
  All three formulations will be transparent solutions. None of the formulations are reported to consistently cause adverse effects at the infusion site. The method of drug administration, including volume and rate of infusion, is identical for all three drugs. These factors ensure that drug administration will be blinded.
  Arms: Levetiracetam

SUMMARY:
The goal of this clinical trial is to determine if treatment of patients with two doses of ketamine plus levetiracetam versus levetiracetam alone leads to more effective control of status epilepticus.

DETAILED DESCRIPTION:
KESETT is a multicenter, randomized, blinded study to determine whether adding 1 mg/kg or 3 mg/kg dose of KET to 60 mg/kg LEV can terminate status epilepticus (SE) in a larger fraction of subjects with benzodiazepine-refractory SE than those treated with LEV (60 mg/kg) alone.

The primary outcome is termination of SE from 15 minutes after starting the study drug infusion, sustained until 60 minutes from enrollment without using additional anti-seizure medication. Termination of SE is determined by (1) improving consciousness and absence of clinically apparent seizures at 60 minutes or (2) absence of any electrographic SE after 15 minutes in those with EEG monitoring and no improvement in consciousness.

Secondary objectives include determining the relative safety of the treatment arms on defined safety outcomes and all adverse events, analysis of secondary/exploratory efficacy outcomes, and evaluation of both effectiveness and safety in the pediatric subpopulation.

The trial will initially allocate subjects equally (1:1:1) for the first 350 participants (burn-in period) before transitioning to response-adaptive randomization. Interim analyses will be conducted for efficacy and futility beginning when 350 subjects have been randomized, and will occur every 100 subjects thereafter. A maximum of 770 participants will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* The patient was witnessed to have a convulsive seizure for greater than 5-minute duration
* The patient received an adequate dose of benzodiazepines. The doses may be divided.
* The last dose of a benzodiazepine was administered 5-30 minutes before study drug administration.
* Continued or recurring seizures in the Emergency Department.
* Age 1 years or older
* Known or estimated weight ≥10 Kg

Exclusion Criteria:

* Known pregnancy
* Prisoner
* Opt-out identification or otherwise known to be previously enrolled in KESETT
* Treatment with a second line anticonvulsant (FOS, PHT, VPA, LEV, phenobarbital, or other agents defined in the MoP) for this episode of SE
* Treatment with sedatives with anticonvulsant properties other than benzodiazepines for this episode of SE(propofol, etomidate, ketamine or other agents defined in the MoP)
* Endotracheal intubation prior to enrollment
* Acute traumatic brain injury clearly precedes seizures
* Scalp injury or burn preventing EEG placement
* Known allergy or other known contraindication to KET or LEV
* Hypoglycemia < 50 mg/dL
* Hyperglycemia > 400 mg/dL
* Cardiac arrest / post-anoxic seizures

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 770 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Termination of SE | From 15 minutes after starting the study drug infusion, sustained for 60 minutes without using additional anti-seizure medication.
  Termination of SE from 15 minutes after starting the study drug infusion, sustained for 60 minutes without using additional anti-seizure medication.
  Termination of SE is determined by (1) improving consciousness and absence of clinically apparent seizures at 60 minutes or (2) absence of any electrographic status epilepticus (ESE) after 15 minutes in those with EEG monitoring and no improvement in consciousness.

SECONDARY OUTCOMES:
Desirability of response (DOOR) outcome | 60 minutes after starting the study drug infusion
  One secondary outcome will be a desirability of response (DOOR) outcome which is a composite efficacy measure evaluated on a graded scale from 1 to 5 at 60 minutes, as follows:
  * No clinically evident or electrographic seizures after 15 minutes, no rescue drugs, and improving mental status by 60 minutes
  * No clinically evident or electrographic seizures after 15 minutes, not intubated, but not improving mental status at 60 minutes
  * No clinically evident or electrographic seizures after 15 minutes, but intubated or use of additional seizures medications (including medications used for intubation)
  * Any clinically evident seizure or electrographic seizure requiring rescue medicine within the timeframe between 15 and 60 minutes
  * Life-threatening hypotension or cardiac arrhythmia or death within 60 minutes
  The Central Adjudication Core will determine the DOOR grade (1-5) based on clinical outcome data provided by the site and EEG data provided by the Central EEG Core.
Endotracheal intubation | Within 60 minutes after start of the study drug infusion
  Endotracheal intubation within 60 minutes of randomization (start of study drug infusion) and duration
ICU duration | Up to 30 days after enrollment
  ICU duration during the study period for those that are admitted to the ICU as abstracted from the hospital admission record
Hospital length-of-stay (LOS) | Up to 30 days after enrollment
  Hospital length-of-stay (LOS) from the ED as abstracted from the hospital admission record
Late recurrent seizure | Between 60 minutes and 4 hours after the start of the study drug infusion
  Number of participants with late recurrent seizure between 60 minutes and 4 hours after the start of the study drug infusion
Time to termination of seizures | From the start of infusion of study drug to the cessation of electrographic seizure assessed up to 60 minutes from study drug initiation
  The interval from the start of infusion of study drug to the cessation of electrographic seizure in those who meet the primary outcome
Late seizures after requiring an anesthetic | Between 60 minutes and 24 hours after start of study drug infusion
  Number of participants with late seizures after requiring an anesthetic between 60 minutes and 24 hours after start of study drug infusion
All cause mortality | From the start of study drug infusion to hospital discharge or day 30
  All cause mortality to end of study

CONTACTS AND LOCATIONS:
Overall Officials: Jaideep Kapur, MD, PhD, Principal Investigator — University of Virginia
Locations (28):
- United States (28):
  - Arthur M. Blank Hospital, Georgia, Alabama
  - Banner University Medical Center - Tucson Campus, Tucson, Arizona
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - Christiana Hospital, Newark, Delaware
  - Nemours Children's Hospital, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Grady Memorial Hospital, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Comer Children's Hospital, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan University Hospital, Ann Arbor, Michigan
  - SUNY Upstate Medical University, Syracuse, New York
  - Duke Regional Hospital, Durham, North Carolina
  - Duke University Hospital, Durham, North Carolina
  - Oregon Health & Science University Hospital, Portland, Oregon
  - Temple University Hospital, Philadelphia, Pennsylvania
  - UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Children's Medical Center Dallas, Dallas, Texas
  - University of Utah Healthcare, Salt Lake City, Utah
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Harborview Medical Center, Seattle, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
The data will be stored in Data Archive for the Brain Initiative (DABI) after trial completion. Once submitted to the data repository, we will work with DABI support to ensure that the de-identified KESETT data is available to the public in the DABI search engine where data requests can be submitted.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The timeline of submission of the public use dataset to the repository will comply with all relevant repository guidelines but in general SIREN will submit data to the repository approximately one year after the primary manuscript of the trial is accepted for publication.
Access Criteria: Access to the de-identified dataset will be controlled by the data repository. DABI offers two approaches to data access: public or private. The KESETT team plans to make the de-identified data public which means it will be publicly available for downloading to DABI account holders.